CLINICAL TRIAL: NCT06189521
Title: Comparison of Extracorporeal Shock Wave Therapy, Ultrasound and Dexamethasone Iontophoresis in Patients With Lateral Epicondylitis
Brief Title: Lateral Epicondylitis Extracorporeal Shock Wave Therapy, Ultrasound Iontophoresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pınar Özge Başaran (Other)
Responsible Party: Sponsor-Investigator, Pınar Özge Başaran, Principal Investigator, Hitit University
Organization: Hitit University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-77
Record Dates: First submitted 2023-12-09; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: This single-blind prospective randomized study. Patients were randomized into three groups by a physiotherapist with sealed envelopes. The researchers were blinded to the patient's groups.
Who Masked: Participant, Care Provider, Investigator
Masking Description: 1. Participant : patients with lateral epicondylitis
  2. Care provider: physiotherapist who applied the treatment (ESWT,US,iontophoresis)
  3. Investigator: examine the patients and evaluates the results of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extracorporeal shock wave group (Active Comparator): Patients were randomized into three groups by a physiotherapist with sealed envelopes. The researchers were blinded to the patient's groups. The same physiotherapy program was applied to all groups. The physiotherapy program consisted of hot packs and TENS for 10 minutes and stretching and eccentric strengthening exercises were given to all groups. All exercises were done under the supervision of the same physiotherapist.
  In addition to the ten-day of physiotherapy program, in the first group one day for a week a total of 3 sessions of ESWT was applied at 1.8 bar, 10.0 Hz, 2000 beats (Elmed Vibrolith Ortho).
  Interventions: Other: Extracorporeal shock wave group
- ultrasound group (Active Comparator): In addition to the ten-day of physiotherapy program, in the second group, ten days of ultrasound applied at 1.5 watt/cm2, continuous mode to the painful area for 5 minutes, 5 days a week for two weeks (Chattanooga Intelect Advanced).
  Interventions: Other: ultrasound group
- dexamethasone iontophoresis group (Active Comparator): In addition to the ten-day of physiotherapy program, in the third group ten days of dexamethasone iontophoresis therapy was applied. 10 days for 10 minutes. 0,1% dexamethasone ophthalmic pomade was applied to the anodal electrode and placed on the lateral epicondyle and 0.1-0.2 milliampere/cm2 galvanic current was applied in each session (ES-522; ITO Physiotherapy and Rehabilitation).
  Interventions: Other: dexamethasone iontophoresis group

INTERVENTIONS:
Other: Extracorporeal shock wave group — In addition to the ten-day of physiotherapy program, in the first group one day for a week a total of 3 sessions of ESWT was applied at 1.8 bar, 10.0 Hz, 2000 beats (Elmed Vibrolith Ortho).
  Arms: Extracorporeal shock wave group
Other: ultrasound group — In addition to the ten-day of physiotherapy program,In the second group, ten days of ultrasound applied at 1.5 watt/cm2 continuous mode to the painful area for 5 minutes, 5 days a week for two weeks (Chattanooga Intelect Advanced).
  Arms: ultrasound group
Other: dexamethasone iontophoresis group — In addition to the ten-day of physiotherapy program, In the third group ten days of dexamethasone iontophoresis therapy was applied. 10 days for 10 minutes. 0,1% dexamethasone ophthalmic pomade was applied to the anodal electrode and placed on the lateral epicondyle and 0.1-0.2 milliampere/cm2 galvanic current was applied in each session (ES-522; ITO Physiotherapy and Rehabilitation).
  Arms: dexamethasone iontophoresis group

SUMMARY:
Lateral epicondylitis (LE) is one of the most common causes of non-traumatic elbow pain, which develops as a result of repetitive stresses due to overuse of the forearm muscles, and is also called tennis elbow.Conservative treatment options include electrotherapy, exercises, extracorporeal shock wave therapy (ESWT), steroid injections, platelet rich plasma, hyaluronic acid injections. As our knowledge this is the first study comparing the three different treatment modalities ESWT, Us and Iontophoresis on lateral epicondylitis The aim of our study; to evaluate the efficacy of ESWT, ultrasound and iontophoresis treatments in terms of pain, grip strength, functionality and quality of life in patients with lateral epicondylitis and to determine the superiority of the treatments against each other.

DETAILED DESCRIPTION:
This is a prospective randomized single blind clinical study. A total of 78 patients age between 18-65 who were diagnosed with lateral epicondylitis between June 2023 and December 2023 were included in our study. The study was approved by the University Ethics Committee (2023-77) and written informed consent was obtained from all the patients. The study was carried out in accordance with the principles of the Declaration of Helsinki.

Patients who had pain at the lateral epicondyle at least for four weeks, detection of sensitivity by palpation on the lateral epicondyle and having positivity in at least two of the special tests (Cozen test, Maudsley test and Mills test) were included in the study. Physical therapy, ESWT or local injections for lateral epicondylitis within the last 3 months, the presence of cervical radiculopathy, carpal tunnel syndrome, other neuropathic diseases, neurologic diseases, medial epicondylitis, systemic inflammatory diseases, tenderness or swelling at the ipsilateral extremity and fibromyalgia have been excluded.

Patients were randomized into three groups by a physiotherapist with sealed envelopes. The researchers were blinded to the patient's groups. The same physiotherapy program was applied to all groups. The physiotherapy program consisted of hot packs and transcutaneus electrical nerve stimulation (TENS) for 10 minutes and stretching and eccentric strengthening exercises were given to all groups. All exercises were done under the supervision of the same physiotherapist.

In addition to the ten-day of physiotherapy program, in the first group one day for a week a total of 3 sessions of ESWT was applied at 1.8 bar, 10.0 Hz, 2000 beats (Elmed Vibrolith Ortho).

In the second group, ten days of ultrasound applied at 1.5 watt/cm2, continuous mode to the painful area for 5 minutes, 5 days a week for two weeks (Chattanooga Intelect Advanced).

In the third group ten days of dexamethasone iontophoresis therapy was applied. 10 days for 10 minutes. 0,1% dexamethasone ophthalmic pomade was applied to the anodal electrode and placed on the lateral epicondyle and 0.1-0.2 milliampere/cm2 galvanic current was applied in each session (ES-522; ITO Physiotherapy and Rehabilitation).

Evaluations were conducted at before treatment and one month after treatment in all groups by the same researchers who were blind in treatment groups.

The clinical and demographic data of the patients were recorded. Numerical Rating Scale (NRS) was used for the pain assessment. The NRS is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). It has been shown that a composite scoring system including best, worse, and current level of pain over the last 24 hours was sufficient to pick up changes in pain intensity with maximal reliability(Jensen et al 1999).

The hand grip strength (HGS) was measured with a Jamar hydraulic hand dynamometer (Saehan, SH5001)) in kilograms. This instrument has a closed hydraulic system that measures the amount of grip strength produced by an isometric contraction applied to the handles and the grip strength of the hand is registered in kilograms Hand and pinch strength were measured by hydraulic pinch gauge (Saehan, SH5005) This instrument has also a closed hydraulic system that measures the amount of grip strength produced by an isometric contraction applied to the handles and the pinc strength of the hand is registered in kilograms Upper extremity disability levels were assessed with Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH). The Quick-DASH is an 11-item that measures upper extremity activity limitation and symptoms . Items were scored from 1: indicating no functional limitation and no symptoms, to 5: indicating functional inability and extreme symptoms. The totalscore was computed by transforming the mean items score to a scale from 0 to 100, where 0 indicates the best upper extremity function and no symptoms. Turkish version of the test was evaluated.

Quality of life was measured by notthingham health profile (NHP). Scale, 6 dimensions, total It consists of 38 items. Sub-dimensions: Energy (3 items), pain (8 items), emotional status (9 items), sleep (5 items),social isolation (5 items) and physical activity (8 items). Its range is 0-100is scored. As the score increases health status gets worse. The validity and reliability of the Turkish version of the test was evaluated.

In the study power analysis performed by examining the related studies in the literature and the sample size required to obtain a significant result was calculated as totally 76 patients, 26 patients in each group (G-Power v3.1.9.7). All data were analysed using the Windows 15.0 Statistical Package for Social Sciences (SPSS Inc., Chicago, IL, USA). Fisher Exact and Chi-square tests were used to determine the differences between proportions or relationships between categorical variables. Paired Sample T-test was used to compare measurements at multiple different times in the same individuals. The Student's t-test was used when the data were normally distributed, the Wilcoxon signed rank test was used for intragroup comparisons and the Mann Whitney U test was used for intergroup comparisons when the data were not normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had pain at the lateral epicondyle at least for four weeks,
* detection of sensitivity by palpation on the lateral epicondyle and
* having positivity in at least two of the special tests (Cozen test, Maudsley test and Mills test) were included in the study

Exclusion Criteria:

* Physical therapy, ESWT or local injections for lateral epicondylitis within the last 3 months,
* the presence of cervical radiculopathy, carpal tunnel syndrome, other neuropathic diseases, neurologic diseases, medial epicondylitis, systemic inflammatory diseases, --
* tenderness or swelling at the ipsilateral extremity and
* patients with fibromyalgia have been excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of ESWT, ultrasound and iontophoresis treatments in term of pain | 6 months from June 2023 to December 2023
  Investigators aimed to evaluate the efficacy of ESWT, ultrasound and iontophoresis treatments in terms of pain, grip strength, functionality and quality of life in patients with lateral epicondylitis.
  Numerical Rating Scale (NRS) was used for the pain assessment The NRS is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Evaluate the efficacy of ESWT, ultrasound and iontophoresis treatments in terms of disability | 6 months from June 2023 to December 2023
  Upper extremity disability levels were assessed with Quick Disabilities of the Arm, Shoulder and Hand questionnaire The Quick-DASH is an 11-item that measures upper extremity activity limitation and symptoms . Items were scored from 1: indicating no functional limitation and no symptoms, to 5: indicating functional inability and extreme symptoms. The tota lscore was computed by transforming the mean items score to a scale from 0 to 100, where 0 indicates the best upper extremity function and no symptoms. Turkish version of the test was evaluated.
  Quality of life was measured by notthingham health profile (NHP) questionaireQuality of life was measured by notthingham health profile (NHP). Scale, 6 dimensions, total It consists of 38 items. Sub-dimensions: Energy (3 items), pain (8 items), emotional status (9 items), sleep (5 items),social isolation (5 items) and physical activity (8 items). Its range is 0-100is scored. As the score increases health status gets worse.

SECONDARY OUTCOMES:
Evaluate the efficacy of ESWT, ultrasound and iontophoresis treatments in terms of strength | 6 months from June 2023 to December 2023
  Investigators aimed to evaluate the efficacy of ESWT, ultrasound and iontophoresis treatments in terms of grip strength, The hand grip strength (HGS) was measured with a Jamar hydraulic hand dynamometer .This instrument has a closed hydraulic system that measures the amount of grip strength produced by an isometric contraction applied to the handles and the grip strength of the hand is registered in kilograms.
  Hand and pinch strength were measured by hydraulic pinch gauge.This instrument has also a closed hydraulic system that measures the amount of grip strength produced by an isometric contraction applied to the handles and the pinc strength of the hand is registered in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: MUSTAFA KESER, MD, Study Chair — HİTİT UNİVERSİTY EROL OLÇOK RESEARCH HOSPİTAL
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No